CLINICAL TRIAL: NCT03276975
Title: A Randomized Trial of CT Fluoroscopy-guided Targeted Autologous Blood and Fibrin Glue Patching for Treatment of Cerebrospinal Fluid Leaks in Spontaneous Intracranial Hypotension.
Brief Title: A Randomized Trial of CT Fluoroscopy-guided Targeted Autologous Blood and Fibrin Glue Patching for Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00083991
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Cerebrospinal Fluid Leaks
Keywords: CT fluoroscopy; epidural patching; spontaneous intracranial hypotension
MeSH Terms: conditions — Cerebrospinal Fluid Leak; Intracranial Hypotension | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patching of CSF Leaks with Autologous Blood and Fibrin (Active Comparator): CT fluoroscopy-guided blood and fibrin glue patching targeted to the site of CSF leak.
  Interventions: Drug: TISSEEL
- Simulated Patching Procedure (Placebo Comparator): Instead of injection of blood and fibrin glue patching material through the needles, an equivalent volume of preservative free sterile Elliots B solution will be injected.
  Interventions: Drug: TISSEEL

INTERVENTIONS:
Drug: TISSEEL — TISSEEL is a fibrin sealant indicated for use as an adjunct to hemostasis in adult and pediatric patients (>1 month of age) undergoing surgery when control of bleeding by conventional surgical techniques (such as suture, ligature, and cautery) is ineffective or impractical. TISSEEL is effective in heparinized patients

SUMMARY:
The goal of this randomized controlled trial (RCT) is to compare the efficacy of CT fluoroscopy-guided targeted epidural patching for treatment of imaging-confirmed spinal CSF leaks to that of a simulated procedure without patching material in patients with spontaneous intracranial hypotension.

DETAILED DESCRIPTION:
Spontaneous intracranial hypotension (SIH) is a condition caused by non-iatrogenic spinal CSF leaks that classically presents with orthostatic headaches. These headaches, in conjunction with other presenting symptoms such as nausea, diplopia, tinnitus, and cognitive deficits, often result in profound disability. SIH is considerably underreported due to pervasive misdiagnosis. Thus, while the estimated annual incidence is reported to be 5 in 100,000, the actual number is likely considerably greater.

The current standard-of-care treatment for SIH cases that are refractory to conservative measures (i.e. bed rest and hydration) is percutaneous epidural blood patching (EBP) of the spinal CSF leak. Percutaneous EBP can be performed in several ways: 1) with or without imaging guidance, 2) targeted to a site of known or suspected CSF leak or non-targeted, and 3) with or without the addition of fibrin glue sealant.

The leading theory for the mechanism behind percutaneous EBP treatment of SIH is that it creates a durable seal of the CSF leak resulting in normalization of CSF hydrodynamics and a resultant diminution in symptoms. Fibrin glue, a sealant used for treatment of unintended durotomies during neurosurgery, is thought to improve the likelihood of a successful patch over patches containing blood alone. Therefore, imaging-guided targeted delivery of patching material containing both blood and fibrin glue directly to the site of CSF leak, a novel therapy, is presumed to be the optimal therapy. For this reason, this procedure has become standard-of-care at many tertiary-care institutions over the past several years.

Our group has extensive experience with CT fluoroscopy-guided targeted blood and fibrin glue patching of proven CSF leaks in SIH patients. However, significant uncertainty remains with regard to the efficacy of this procedure due to a paucity of outcomes data and the absence of any prospective RCTs. In fact, nearly all of the current evidence for the treatment of SIH is found in the form of retrospective chart reviews. Given the growing recognition of SIH, the fact that a known subset of patients will have spontaneous resolution of symptoms, and the absence of clear evidence to guide treatment, there is a critical need to evaluate the efficacy of targeted patching with blood and fibrin glue with a prospective RCT. Fulfilling this unmet need forms the basis for this proposal. While determining the efficacy of the other types of EBPs is also important, we aim to begin by evaluating the efficacy of the presumed optimal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients meeting International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria for a diagnosis of SIH (Table 1) who have had a contrast-enhanced brain MRI and a myelogram confirming the presence of a CSF leak will be recruited from the Duke Radiology spine intervention clinic [25]

Exclusion Criteria:

* recent (i.e., < 2 weeks) blood patch
* contraindication or inability to undergo the procedure
* inability to provide informed consent
* expected inability to complete follow-up assessment
* a contraindication to receiving contrast material (precluding an epidurogram)
* contraindication to receiving fibrin glue (i.e., allergy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue: CT-fluoroscopic guided epidural patching of the CSF leak or CSF to venous fistula with autologous blood and fibrin glue.
- Simulated Patching Procedure: A simulated procedure in which CT fluoroscopy is used to place needles but instead of injection of blood and fibrin glue patching material, an equivalent volume of preservative free sterile saline is injected.
Period: Overall Study
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
Started | 8 | 7
Crossover At 2 Months | 0 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.1) | 57.6 (14.7) | 51.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 3 | 4 | 7
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Median (Headache Impact Test-6) HIT-6 Score From Baseline
Description: Absolute change in median HIT-6 score from pre-procedural baseline to 1 month post procedure for each group. The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often", or "always". These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent.
Time Frame: Baseline, 1 month
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
Number analyzed (Participants) | 8 | 7
score on a scale | -12 [-16 to -7] | -7 [-13 to -1]

2. Secondary Outcome: Change in Median HIT-6 Score From Baseline
Description: Absolute change in median HIT-6 score from pre-procedural baseline to 2 weeks and 4 months post procedure for each group. The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often", or "always". These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent.
Time Frame: Baseline, 2 weeks, 4 months
Population: All patients at the 4 month time point in the Simulated Patching Procedure Arm/Group had crossed over to the Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue Arm/Group
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
Number analyzed (Participants) | 8 | 7
units on a scale
  2 weeks | -5.5 [-10 to 0.5] | -7 [-17 to -3]
  4 months | -4.5 [-16.5 to -1.5] | -12 [-24 to -7]

3. Secondary Outcome: Reduction in Median Migraine Disability Assessment (MIDAS) Score From Baseline
Description: The MIDAS questionnaire assesses headache-related disability. Patients answer five questions, scoring the number of days, in the past 3 months, where their activity was limited due to headache. A higher score indicates greater headache-related disability. This tool has been shown to be internally consistent, highly reliable, valid, and correlates with physicians' clinical judgment. MIDAS Scale Range: 0 - 270
Time Frame: Baseline, 2 weeks, 1 month, 4 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
Number analyzed (Participants) | 8 | 7
units on a scale
  2 weeks | -25 [-55 to 6] | 16 [-35 to 100]
  1 month | -62.5 [-117 to -37] | -40 [-86 to -3]
  4 months | -87 [-134.5 to -69.5] | -53 [-210 to -22]

4. Secondary Outcome: Change in Median NRS Score From Baseline
Description: The pain numerical rating scale (NRS) is a well-validated tool for quantitatively assessing patients' pain. The NRS asks patients to rate their current pain intensity on an 11-point scale ranging from 0 ("no pain") to 10 ("worst possible pain"). It has been found to be a valid measure of pain intensity with minimum clinically important difference noted to be a change of 2 points. The investigators will use NRS averaged over the past 24 hours for all time points in this trial. The Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consensus statement indicates that an NRS reduction of 30% (or 2 points) is associated with a meaningful or moderately important improvement in pain. Further, IMMPACT also indicates that an NRS reduction of 50% (or 4 points) is associated with a substantial improvement in pain. The investigators will follow their consensus recommendations and explicitly report these two categories of pain relief.
Time Frame: Baseline, 2 weeks, 1 month, 4 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
Number analyzed (Participants) | 8 | 7
units on a scale
  2 weeks | -0.5 [-1.5 to 1] | -1 [-3 to 0]
  1 month | -2.5 [-4.5 to -1] | 0 [-3 to 3]
  4 months | -1.5 [-5 to -0.5] | -2 [-3 to -1]

5. Secondary Outcome: Change in Median EQ-5D (European Quality of Life-5 Dimensions) Score From Baseline
Description: The EQ-5D is a standardized measure of health status that provides a simple, generic measure of health for clinical appraisal. It is well-validated for health status measurement and for quality-of-life in headache. Scores on the EQ-5D were calculated using the United States 3L, time trade off (TTO) valuation technique. Scores range from 0 to 1, with 1 indicating perfect health.
Time Frame: Baseline, 2 weeks, 1 month, 4 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
Number analyzed (Participants) | 8 | 7
units on a scale
  2 weeks | 0.1 [0 to 0.2] | 0.1 [-0.1 to 0.3]
  1 month | 0 [0 to 0.4] | 0.1 [0 to 0.4]
  4 months | 0 [-0.1 to 0.1] | 0.2 [0.1 to 0.4]

6. Secondary Outcome: Change in Median WPAI (Work Productivity and Activity Impairment) Score From Baseline
Description: The WPAI is a validated instrument with good test-retest reliability used extensively in health research that quantifies impairment in daily activities and work productivity. Scores on the WPAI range from 0 - 100% with higher percentages indicating greater impact on work productivity and more severe activity impairment.
Time Frame: Baseline, 2 weeks, 1 month, 4 months
Population: Patients were only analyzed with respect to WPAI if they were currently employed at the time of the outcome measure acquisition (for each time point). Thus, there were fewer patients for whom data was recorded than were enrolled in each arm (number analyzed).
  All patients at the 4 month time point in the Simulated Patching Procedure Arm/Group had crossed over to the Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue Arm/Group
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
Number analyzed (Participants) | 8 | 7
units on a scale
  2 weeks: number analyzed (Participants) | 8 | 4
  2 weeks | 1.3 [-16.9 to 13.5] | -0.3 [-8.8 to 3.6]
  1 month: number analyzed (Participants) | 8 | 4
  1 month | -13.8 [-51 to 5] | -2.3 [-20.8 to 20]
  4 months: number analyzed (Participants) | 7 | 2
  4 months | -9 [-29 to 13.7] | -28.5 [-47 to -10]

7. Secondary Outcome: Change in PGIC (Patient Global Impression of Change) Score From Baseline
Description: PGIC is a validated 7-point Likert-type scale assessing a patient's overall impression of improvement after intervention. Scores range from 1 - 7 (1: no change or worsening of condition; 2: almost the same, hardly any change at all; 3: a little better, but no noticeable change; 4: somewhat better, but the change has not made any real difference; 5: moderately better, and a slight but noticeable change; 6: better and a definite improvement that has made a real and worthwhile difference; 7: a great deal better, and a considerable improvement that has made all the difference) with higher scores indicating greater improvement.
Time Frame: Baseline, 2 weeks, 1 month, 4 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
Number analyzed (Participants) | 8 | 7
score on a scale
  2 weeks | 3.5 [3 to 4.5] | 2 [1 to 4]
  1 month | 4 [3 to 5.5] | 3 [1 to 5]
  4 months | 4.5 [3.5 to 6] | 6 [2 to 6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected immediately after the initial procedure, immediately after any crossover procedures (performed at the 2-month time point), and also at 1 week after any procedure (initial or crossover).
Description: All 7 participants in the Simulated Patching Procedure arm chose to cross over to the Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue arm at the 2-month time point. Therefore, a total of 15 participants received the Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue intervention.
Arm/Group | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue | Simulated Patching Procedure
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/7
Other Adverse Events (participants affected / at risk) | 1/15 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted Epidural Patching of CSF Leaks With Autologous Blood and Fibrin Glue (N=15) | Simulated Patching Procedure (N=7)
Asymptomatic self-limited hypertension (Vascular disorders) | 0 (0) | 1 (1) — Patient had mild asymptomatic self-limited hypertension while in the recovery room. No untoward effects. Discharged in good condition.
Rebound Intracranial Hypertension (Nervous system disorders) | 1 (1) | 0 (0) — Patient experience a headache of new phenotype after the procedure that was self-limited and consistent with rebound intracranial hypertension, a known and expected event after patching procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT03276975/Prot_SAP_000.pdf